CLINICAL TRIAL: NCT01289600
Title: The Role of Diaphragm Electromyography (EMG) Guided Mechanical Ventilation on Respiratory Physiology in Mechanically Ventilated Patients With Acute Respiratory Distress Syndrome (ARDS)
Brief Title: Mechanical Ventilation and Respiratory Muscle Work of Breathing in Acute Respiratory Distress Syndrome (ARDS) Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Nijmegen (Other)
Responsible Party: Principal Investigator, Leo Heunks, MD PhD, University Medical Center Nijmegen
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ARDS1
Record Dates: First submitted 2011-01-27; First posted 2011-02-04 (Estimated); Last update posted 2015-06-10 (Estimated); Status verified 2015-06

CONDITIONS: ARDS
MeSH Terms: interventions — Respiration, Artificial

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Pressure support ventilation, ARDSnet (Active Comparator): Mechanical ventilator is set to pressure support ventilation (6 ml/kg) for 30 min with positive end expiratory pressure (PEEP) set according to the "higher arm" of the ARDS network consensus.
  Interventions: Device: Mechanical ventilation
- Pressure control ventilation, ARDSnet (Active Comparator): Mechanical ventilator is set to pressure control ventilation (6 ml/kg) for 30 min with PEEP set according to the "higher arm" of the ARDS network consensus.
  Interventions: Device: Mechanical ventilation
- Neurally adjusted ventilatory assist, ARDSnet (Active Comparator): Mechanical ventilator is set to NAVA for 30 min with PEEP set according to the "higher arm" of the ARDS network consensus.
  Interventions: Device: Mechanical ventilation
- Neurally adjusted ventilatory assist, titrated (Active Comparator): Mechanical ventilator is set to NAVA for 30 min with PEEP titrated using the diaphragm EMG signal.
  Interventions: Device: Mechanical ventilation

INTERVENTIONS:
Device: Mechanical ventilation — The mechanical ventilator is set to different ventilation modes as described in the individual arms.
  Other Names: Maquet Servo-i

SUMMARY:
The purpose of this study is to demonstrate that mechanical ventilation guided by the diaphragm EMG signal (also know as neurally adjusted ventilatory assist [NAVA]) is superior compared to pressure support and pressure control ventilation.

ELIGIBILITY:
Inclusion Criteria:

* intubated, mechanically ventilated patients
* meeting criteria for ARDS
* mean arterial blood pressure > 65 mmHg (with or w/o vasopressors)

Exclusion Criteria:

* pregnancy
* increased intracranial pressure
* contra-indication naso-gastric tube
* diagnosed neuro-muscular disorder
* recent (<12 hours) use of muscle relaxants
* exclusion from sedation interruption protocol as used in our institution
* open chest or- abdomen
* very high inspiratory flow rate during supported ventilation
* inability to obtain informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2011-01; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Pressure-time product of the diaphragm | average of last 15 minutes of each study arm
  The pressure-time product of the transdiaphragmatic pressure (Pdi) during inspiration is obtained for each breath by multiplying the corresponding mean inspiratory Pdi signal above the end-expiratory baseline by the inspiration time. Breath-by-breath data are ensemble-averaged over the last 15 minutes of each study arm.
Patient - ventilator asynchrony index | average of last 15 minutes of each study arm
  Ventilator asynchrony is determined as the sum of the triggering and cycling-off delays per breath, expressed as a percentage of the total breath duration. The trigger delay is measured as the time difference between the onset of neural inspiration and the ventilator inspiratory flow, and the cycling delay as the time difference between the end of neural inspiration and the end of ventilator inspiratory flow. Breath-by-breath data are ensemble-averaged over the last 15 minutes of each study arm.

SECONDARY OUTCOMES:
Transpulmonary pressure | average of last 15 minutes of each study arm
  Transpulmonary pressure is determined as the difference between mouth pressure and esophageal pressure during inspiration. Breath-by-breath data are ensemble-averaged over the last 15 minutes of each study arm.
Transdiaphragmatic pressure | average of last 15 minutes of each study arm
  Transdiaphragmatic pressure is determined as the difference between gastric pressure and esophageal pressure during inspiration. Breath-by-breath data are ensemble-averaged over the last 15 minutes of each study arm.
Oxygenation index | at the end of each study arm
  Oxygenation index is determined as the ratio between arterial oxygen tension and fraction of inspired oxygen. Arterial oxygen tension is obtained at the end of each study arm.
Dead space ventilation | average of last 15 minutes of each study arm
  Dead space ventilation is determined each breath using the Bohr equation: (PaCO2-PeCO2/PaCO2)*Vt. Here Vt is tidal volume, PaCO2 is the partial pressure of carbon dioxide in the arterial blood, and PeCO2 is the end-tidal carbon dioxide tension in the expired air. Breath-by-breath data are ensemble-averaged over the last 15 minutes of each study arm.

CONTACTS AND LOCATIONS:
Overall Officials: Leo Heunks, MD, PhD, Principal Investigator — Radboud University Nijmegen Medical Center
Locations (1):
- University Medical Center Nijmegen, Nijmegen, Gelderland, Netherlands